CLINICAL TRIAL: NCT06434376
Title: Study on Adjuvant Treatment of MRD-positive Colorectal Cancer Patients With Routine Chemotherapy Combined With Personalized Immune Regulation Diagnosis and Treatment Technology
Brief Title: MRD-positive Colorectal Cancer Patients Combined With Personalized Immune Regulation Diagnosis
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAHoWMU-CR2024-02-110
Record Dates: First submitted 2024-05-23; First posted 2024-05-30 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-04

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): Conventional adjuvant therapy combined with personalized immune regulation diagnosis and treatment technology
  Interventions: Biological: Conventional chemotherapy combined with personalized immune regulation diagnosis and treatment technology

INTERVENTIONS:
Biological: Conventional chemotherapy combined with personalized immune regulation diagnosis and treatment technology — Blood samples were collected for MRD detection within one month (week 3) after colorectal cancer surgery, and MRD-positive patients were selected for routine chemotherapy (course of 6 months). Blood and tumor tissue samples of enrolled patients were collected, and relevant clinical data were recorded. The whole exon and expression profile of surgical tumor tissue samples were sequenced, neoantigens were analyzed, and immunomodulators were prepared. After the preparation of individualized immunomodulators, combined treatment was performed simultaneously with chemotherapy. During the treatment process, patients' response to treatment and survival were observed, and tumor load, ctDNA changes, imaging and other indicators before and after treatment were compared. To evaluate the efficacy of immunotherapy.

SUMMARY:
Establish the clinical technology system of routine adjuvant therapy combined with personalized immune regulation diagnosis and treatment technology for postoperative anti-relapse adjuvant therapy: Patients with MRD positive and high risk of recurrence after colorectal cancer surgery were enrolled. Surgical tumor tissue and blood samples were collected, tumor tissue samples were sequenced, neoantigens were analyzed, personalized immunomodulators were prepared, and routine adjuvant therapy combined with personalized immunomodulatory diagnosis and treatment technology were performed to prevent postoperative recurrence. To establish the clinical technology system of routine adjuvant therapy combined with personalized immune regulation diagnosis and treatment technology for postoperative anti-relapse adjuvant therapy

ELIGIBILITY:
Inclusion Criteria:

1. They must give informed consent, indicating that they understand the purpose of the study and the procedures required, and are willing to participate in the study.
2. Age 18-80.
3. Pathological examination confirmed colorectal adenocarcinoma.
4. For patients with stage II with high risk factors or stage III with radical surgery, stage II (high risk) colon cancer is defined as (any of):

   a )T4 b)≥ Level 3 c) The clinical manifestations are intestinal obstruction or intestinal perforation d) Histological signs of vascular, lymphatic, or perineural invasion e) Check < 12 nodes
5. Patients with liver or lung metastases that can be resected in one stage with the primary lesion.
6. There must be sufficient formalin to fix the tumor material in the paraffin embedded (FFPE) block or section tissue (only after sponsor approval), preferably obtained from excision.
7. Patients should meet the following biochemical indicators: total bilirubin ≤2× upper limit of normal (ULN); AST and ALT≤2× upper limit of normal (ULN); Creatinine clearance ≥60 ml/min.
8. Patients should meet the following hematological indicators: neutrophil count ≥1.5×109 /L; Hemoglobin ≥10.0 g/dL; Platelet count ≥100×109 /L.
9. Expected survival ≥ 3 months.
10. Postoperative ctDNA MRD test was positive, routine blood indexes were negative, and imaging was negative.

Exclusion Criteria:

1. Stage I patients and stage II patients without risk factors or MSI-H.
2. Stage IV patients who cannot be surgically resected.
3. Patients with liver, kidney, heart, lung and other dysfunction, unable to tolerate surgery or unable to complete follow-up chemotherapy.
4. Patients who refuse adjuvant therapy such as chemotherapy, are allergic to chemotherapy drugs and have poor compliance.
5. Patients who have received other immunotherapy within 1 month (such as immune checkpoint inhibitor therapy, therapeutic antibody therapy, immune cell therapy, and immune system modulator therapy)
6. Patients with a known past or current malignancy, except where a diagnosis is included, except in the following cases:

   1. Stage 1B or below cervical cancer.
   2. Non-invasive basal cell or squamous cell skin cancer.
   3. Non-invasive superficial bladder cancer.
   4. Prostate cancer with a current PSA level < 0.1 ng/mL.
   5. Any curable cancer with a complete response (CR) duration of > 2 years.
7. Patients with hematological and autoimmune diseases.
8. Patients with active hepatitis B or C.
9. Patients affected by drug abuse, clinical or psychological or social factors that make informed consent or the implementation of research.
10. Pregnant and lactating women.
11. Patients with mental illness, senile dementia, etc.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2024-07-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
ORR | Visits were conducted at the end (or termination) of each course and at 30, 90, and 120 days after the end of the last course for 4 months
  Exploration of the efficacy of Conventional adjuvant therapy combined with personalized immune regulation diagnosis and treatment technology

SECONDARY OUTCOMES:
PFS | Visits were conducted at the end (or termination) of each course and at 30, 90, and 120 days after the end of the last course for 4 months
  Observe and evaluate the progression free survival (PFS) of Postoperative MRD positive patients with with routine chemotherapy combined with personalized immune regulation diagnosis and treatment technolog
OS | Visits were conducted at the end (or termination) of each course and at 30, 90, and 120 days after the end of the last course for 4 months
  Observe and evaluate the overall survival(OS) of Postoperative MRD positive patients with with routine chemotherapy combined with personalized immune regulation diagnosis and treatment technology

IPD SHARING:
Plan to Share IPD: No
publication